CLINICAL TRIAL: NCT05405894
Title: Efficacy of a Single Infusion of Zoledronic Acid to Mitigate the Rebound Effect of Rapid Bone Loss Following Denosumab Treatment Discontinuation
Brief Title: Efficacy of Zoledronic Acid to Prevent Bone Loss Following Denosumab Discontinuation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB21-1898
Record Dates: First submitted 2022-05-27; First posted 2022-06-06 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-11

CONDITIONS: Osteoporosis; Osteoporosis, Postmenopausal; Osteopenia; Bone Loss
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal; Bone Diseases, Metabolic | interventions — Zoledronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Zoledronic acid — Once-yearly infusion of zoledronic acid following denosumab discontinuation
  Other Names: Dr. Reddy's Zoledronic acid

SUMMARY:
This two-year observational, open-label clinical trial will evaluate the efficacy of a once-yearly infusion of zoledronic acid after denosumab discontinuation to maintain tissue mineral density and bone microarchitecture using high-resolution peripheral quantitative computed tomography (HR-pQCT) among post-menopausal women with osteoporosis.

DETAILED DESCRIPTION:
As part of an observational study, twenty female osteoporosis patients looking to transition off denosumab therapy will be recruited from the David Hanley Osteoporosis Centre and affiliated primary care physicians in Calgary. The decision to stop denosumab will be made in accordance with standard clinical care and fully separate from the present study. Approximately 6-8 months after the patients' final denosumab injection, patients will receive a single infusion of zoledronic acid (5 mg/100mL) as part of their routine standard of care. The 6-8 month time frame corresponds with the recommended duration between subsequent denosumab injections. Concurrent with zoledronic acid treatment (within one month before or after infusion), patients will visit to the McCaig Institute for Bone and Joint Health to receive a baseline dual X-ray absorptiometry scan (lumbar spine, lateral vertebral assessment, and hip) and a high-resolution peripheral computed tomography scan (radius and tibia) to quantify areal BMD and volumetric BMD/bone microarchitecture, respectively. They will also complete the MoJo Fracture Risk Questionnaire. Patients will return for repeat scanning and questionnaire administrations to monitor potential changes to bone at 6 and 12 months after baseline. Any fracture events during the 12-month time frame will be logged in consultation with the patients' physician as documented through routine clinical follow-up. Researchers may contact participants to repeat scanning and questionnaire administration at the 24-month time point, if participants agree to this contact within the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal females with osteoporosis
* Anticipating or preparing to transition off active denosumab treatment for osteoporosis with the use of a once-yearly infusion of zoledronic acid
* Received at least 2 injections of denosumab treatment
* Had a recent test (within 6 months) of serum creatine, calcium and phosphate

Exclusion Criteria:

* Any person for whom zoledronic acid would be considered contraindicated
* Pre-menopausal females
* Any person with significant chronic kidney disease (eGFR < 50 ml/m2 at time of osteoporosis clinical assessment)
* Any person with previous adverse reactions or allergy to bisphosphonate therapies
* Any person with non-corrected hypocalcaemia
* Any person currently taking, and unable to discontinue the use of, prohibited medications including: ZOMETA, other bisphosphonate therapies, calcitonin, aminoglycosides, loop diuretics and agiogenesis inhibitors
* Any person with other history, condition, therapy, or uncontrolled intercurrent illness, which could in the opinion of the Qualified Medical Investigator affect compliance with study requirements or which would make the participant unsuitable for this study
* Any person with simultaneous participation in another interventional clinical study (e.g., Phase 1-3 clinical studies) or treatment with any investigational medicinal product within 30 days prior to screening visit

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study focuses on post-menopausal, osteoporotic females, anticipating or preparing to transition off active denosumab treatment, for which they have received at least 2 prior injections, via a transition to once-yearly infusion of zoledronic acid.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in volumetric Bone Mineral Density (BMD)/bone microarchitecture from baseline | Change from Baseline (within 1-month of infusion) to 6-months and 12-months
  High-resolution peripheral computed tomography scan (radius and tibia) will be used to quantify volumetric BMD/bone microarchitecture
Change in areal Bone Mineral Density (BMD) from baseline | Change from Baseline (within 1-month of infusion) to 6-months and 12-months
  Dual X-ray absorptiometry scan (lumbar spine, lateral vertebral assessment, and hip) will be used to quantify areal BMD

SECONDARY OUTCOMES:
Fractures | 1 year
  Any clinically diagnosed fractures will be reported by treating physician
MoJo Fracture Risk Questionnaire | 1 year
  An assessment of fracture risk

OTHER OUTCOMES:
Optional further assessment of change in volumetric Bone Mineral Density (BMD)/bone microarchitecture from baseline | Change from Baseline to 24-months
  High-resolution peripheral computed tomography scan (radius and tibia) will be used to quantify volumetric BMD/bone microarchitecture
Optional further assessment of change in areal Bone Mineral Density (BMD) from baseline | Change from Baseline to 24-months
  Dual X-ray absorptiometry scan (lumbar spine, lateral vertebral assessment, and hip) will be used to quantify areal BMD

CONTACTS AND LOCATIONS:
Overall Officials: William Brent Edwards, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, McCaig Institute for Bone and Joint Health, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solling AS, Harslof T, Langdahl B. Treatment with Zoledronate Subsequent to Denosumab in Osteoporosis: a Randomized Trial. J Bone Miner Res. 2020 Oct;35(10):1858-1870. doi: 10.1002/jbmr.4098. Epub 2020 Jul 12. PMID 32459005
- [Background] Anastasilakis AD, Polyzos SA, Makras P, Aubry-Rozier B, Kaouri S, Lamy O. Clinical Features of 24 Patients With Rebound-Associated Vertebral Fractures After Denosumab Discontinuation: Systematic Review and Additional Cases. J Bone Miner Res. 2017 Jun;32(6):1291-1296. doi: 10.1002/jbmr.3110. Epub 2017 Mar 13. PMID 28240371